CLINICAL TRIAL: NCT00383331
Title: A Phase II Study of ALIMTA® (Pemetrexed) and GEMZAR® (Gemcitabine) Every 14 Days Versus Pemetrexed and Gemcitabine Every 21 Days in Advanced Non-Small Cell Lung Cancer
Brief Title: Pemetrexed and Gemcitabine Every 14 Days Versus Every 21 Days in Advanced Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was stopped early due to low enrollment
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9431; H3E-US-S061
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2009-05-14 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-05

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Gemcitabine
- B (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed — A: 500 mg/m2, intravenous (IV), every 21 days x 6 cycles
  B: 500 mg/m2, intravenous (IV), every 14 days x 9 cycles
  Other Names: LY231514; Alimta
Drug: Gemcitabine — A: 1250 mg/m2, intravenous (IV) days 1 and 8, every 21 days x 6 cycles
  B: 1500 mg/m2, intravenous (IV), every 14 days x 9 cycles
  Other Names: LY188011; Gemzar

SUMMARY:
This study is designed to evaluate Pemetrexed and Gemcitabine Day 1 followed by Gemcitabine Day 8 every 21 days (Arm A) and Pemetrexed and Gemcitabine Day 1 every 14 days (Arm B) in patients with NSCLC. Each agent and sequence has well demonstrated antitumor activity respectively in patients with locally advanced or metastatic NSCLC. Therefore, it is reasonable to investigate the most optimal schedule for this combination, and which combination is associated with the most anti-tumor activity in the phase II arena.

ELIGIBILITY:
Inclusion Criteria:

* histologic or cytologic diagnosis of NSCLC Stage IIIB or IV
* no prior systemic chemotherapy for advanced Non-Small Cell Lung Cancer
* Prior radiotherapy must be completed at least 4 weeks before study enrollment.

Exclusion Criteria:

* estimated life expectancy of 12 weeks
* a serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease
* documented brain metastases unless the patient has completed successful local therapy for central nervous system metastases and has been off of corticosteroids for at least 2 weeks before enrollment
* significant weight loss (that is, > 10%) over the previous 6 weeks before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 21-Day Cycle: Pemetrexed and Gemcitabine Day 1 followed by Gemcitabine Day 8, every 21 days x 6 cycles
- 14-Day Cycle: Pemetrexed and Gemcitabine Day 1, every 14 days x 9 cycles
Period: Overall Study
Arm/Group | 21-Day Cycle | 14-Day Cycle
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 21-Day Cycle | 14-Day Cycle | Total
Number analyzed (Participants) | 10 | 9 | 19
Age Continuous [Median (Full Range); unit: years] | 70.5 [60.0 to 81.0] | 63.0 [48.0 to 74.0] | 66.0 [48.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
Eastern Cooperative Oncology Group Performance Score [Number; unit: participants]
  0 - Fully Active | 4 | 4 | 8
  1 - Ambulatory, Restricted Strenuous Activity | 6 | 5 | 11
  2 - Amublatory, No Work Activities | 0 | 0 | 0
  3 - Partially Confined to Bed, Limited Self Care | 0 | 0 | 0
  4 - Completely Disabled | 0 | 0 | 0
Previous Radiation Therapy [Number; unit: participants]
  Yes | 3 | 1 | 4
  No | 7 | 8 | 15
Stage of Lung Cancer [Number; unit: participants]
  IIIB with pleural effusion | 2 | 2 | 4
  IV | 8 | 7 | 15
Tumor Cell Type [Number; unit: participants]
  Squamous | 1 | 2 | 3
  Adenocarcinoma | 5 | 3 | 8
  Non-Small Cell Lung, Not Otherwise Specified (NOS) | 4 | 2 | 6
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment.
Time Frame: baseline and every 14 or 21 day cycle (6-9 cycles), every 6 weeks post-therapy follow-up
Measure: Number; unit: participants
Arm/Group | 21-Day Cycle | 14-Day Cycle
Number analyzed (Participants) | 10 | 8
participants
  Complete Response | 0 | 0
  Partial Response | 2 | 0
Statistical Analysis 1: Comparison: 21-Day Cycle vs 14-Day Cycle; The response rates are separately evaluated for these two treatment arms. For each arm, a sample size of 48 achieves 91% power to detect a difference of 20% between the null hypothesis of 15% response rate and the alternative hypothesis of 35% using a one-sided, binomial hypothesis test with a target significance level of 2.5% (the actual significance level is 2.2%); Test type: Superiority or Other; p = 0.48, Fisher Exact

2. Secondary Outcome: Progression Free Survival
Description: baseline to measured progressive disease
Time Frame: baseline and every 14 or 21 day cycle (6-9 cycles), every 6 weeks post-therapy follow-up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 21-Day Cycle | 14-Day Cycle
Number analyzed (Participants) | 10 | 8
months | 1.66 [0.69 to 4.30] | 5.04 [1.74 to 5.95]

3. Secondary Outcome: Time to Progressive Disease
Description: Time to progressive disease not analyzed because trial was stopped early due to low enrollment.
Time Frame: baseline and every 14 or 21 day cycle (6-9 cycles), every 6 weeks post-therapy follow-up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 21-Day Cycle | 14-Day Cycle
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response
Description: Duration of response was not analyzed because the trial was stopped early due to low enrollment.
Time Frame: baseline and every 14 or 21 day cycle (6-9 cycles), every 6 weeks post-therapy follow-up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 21-Day Cycle | 14-Day Cycle
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was not analyzed because the trial was stopped early due to low enrollment.
Time Frame: baseline and every 14 or 21 day cycle (6-9 cycles), every 6 weeks post-therapy follow-up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 21-Day Cycle | 14-Day Cycle
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival
Description: Survival time is defined as the time from date of randomization to death due to any cause.
Time Frame: baseline and every 14 or 21 day cycle (6-9 cycles), every 6 weeks post-therapy follow-up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 21-Day Cycle | 14-Day Cycle
Number analyzed (Participants) | 10 | 8
months | 5.1 [2.4 to 14.2] | 8.1 [5.5 to 10.1]
Statistical Analysis 1: Comparison: 21-Day Cycle vs 14-Day Cycle; Test type: Superiority or Other; p = 0.56, Log Rank

ADVERSE EVENTS:
Arm/Group | 21-Day Cycle | 14-Day Cycle
Serious Adverse Events (participants affected / at risk) | 9 | 4
Other Adverse Events (participants affected / at risk) | 10 | 9
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | 21-Day Cycle | 14-Day Cycle
Thrombocytopenia (Blood and lymphatic system disorders) | 1/10 (1) | 0/9 (0)
Ischemia-Cerebral (Nervous system disorders) | 1/10 (1) | 0/9 (0)
Disease Progression - Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/10 (2) | 0/9 (0)
Fatigue (General disorders) | 0/10 (0) | 2/9 (2)
Neutropenia (Blood and lymphatic system disorders) | 2/10 (2) | 2/9 (2)
Leukopenia (Blood and lymphatic system disorders) | 1/10 (1) | 0/9 (0)
Pain - Extremity (General disorders) | 1/10 (1) | 0/9 (0)
Anemia (Blood and lymphatic system disorders) | 1/10 (1) | 0/9 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 15% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | 21-Day Cycle | 14-Day Cycle
Nausea (Gastrointestinal disorders) | 5/10 | 7/9
Thrombocytopenia (Blood and lymphatic system disorders) | 7/10 | 2/9
Diarrhea-No Colostom (Gastrointestinal disorders) | 4/10 | 2/9
Anorexia (Psychiatric disorders) | 2/10 | 3/9
Constipation (Gastrointestinal disorders) | 3/10 | 1/9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2/10 | 2/9
Pneumonia NOS (Respiratory, thoracic and mediastinal disorders) | 0/10 | 4/9
Pruritis (Infections and infestations) | 3/10 | 1/9
Rash (Skin and subcutaneous tissue disorders) | 3/10 | 1/9
Vomiting (Gastrointestinal disorders) | 2/10 | 2/9
Anemia (Blood and lymphatic system disorders) | 8/10 | 8/9
Leukopenia (Blood and lymphatic system disorders) | 8/10 | 8/9
Neutropenia (Blood and lymphatic system disorders) | 6/10 | 6/9
Fatigue (General disorders) | 6/10 | 4/9

LIMITATIONS AND CAVEATS:
Trial was stopped early due to low enrollment. Some secondary outcomes were not analyzed due to the low numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days